CLINICAL TRIAL: NCT07371832
Title: A Single Center Evaluation of AI Enabled SureForm Robotic Stapler (SureformTM) Compared to Conventional Stapler for Colorectal Cancer Procedures
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterology, Asian Institute of Gastroenterology, India
Other Study IDs: STAPLER
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic-Assisted Surgery Group (Intervention Arm): Subjects undergoing robotic-assisted colorectal cancer surgery where AI-enabled SureForm™ Robotic.Stapler is used for bowel transection and/or creation of anastomosis.
  Interventions: Device: AI-enabled SureForm™ Robotic Stapler; Device: Conventional Laparoscopic Stapler
- Laparoscopic Surgery Group (Comparator Arm): Subjects undergoing laparoscopic colorectal cancer surgery using conventional laparoscopic staplers for bowel transection and/or creation of anastomosis.
  Interventions: Device: AI-enabled SureForm™ Robotic Stapler; Device: Conventional Laparoscopic Stapler

INTERVENTIONS:
Device: AI-enabled SureForm™ Robotic Stapler — Use of AI-enabled SureForm™ robotic stapler during robotic-assisted colorectal resections for transection and/or anastomosis creation.
Device: Conventional Laparoscopic Stapler — Use of standard conventional laparoscopic staplers during laparoscopic colorectal resections for transection and/or anastomosis creation

SUMMARY:
Robotic-assisted surgeries are especially valuable for colorectal pathologies because they offer better vision and control for surgical manipulation given the narrow operative region within the pelvis .Some of the iatrogenic risk factors associated with higher post-operative adverse events following colorectal surgeries are surgeon experience' and hospital case load'. In order to mitigate these factors, surgical staplers have gained preference amongst surgeons due to their reproducible results and ease of learning At present there are only two methods of creating an anastomosis: hand-sewn technique using sutures or surgical staplers. Surgical staplers have been shown to be as effective as hand-sewn techniques for colorectal anastomoses However, anastomotic strictures can be bothersome for patients and the rate of stricture is fourfold higher for stapled anastomoses than for those that are hand sewn in colorectal anastomoses . Additionally, overzealous or incorrect stapling could also result in hemostasis or ischemia One of the most dreaded adverse events of colorectal resection is anastomotic leakages followed, in decreasing severity, by post-operative bleeding and ileus. Because of the severity of adverse events associated with an anastomotic leak, it is important to detect it early and provide early management for the same. However, diagnosis of anastomotic leakage is commonly a symptomatic diagnosis based on development of gas, purulent or fecal discharge from the drain, purulent discharge from the rectum, pelvic abscess or peritonitis. Such severe symptoms further complicate the post-operative recovery and lengthen the hospital stay. Interestingly, it has been

reported that anastomotic leaks were more often diagnosed late in the postoperative period and more often after hospital discharge, or 12 days postoperatively . Anastomotic leakage rates vary from the colon to the rectum, with much higher rates in the rectum. Because of the severity of adverse events associate with an anastomotic leak, there is a pressing need for new techniques for prevention of anastomotic leakages .

ELIGIBILITY:
Inclusion Criteria:

A. Subjects, 18 to 90 years B. Subjects who will undergo Planned robotic-assisted surgery or laparoscopic surgery (as the primary treatment) for non-metastatic colorectal cancer where staplers are utilized for transection and/or creation of anastomosis

Exclusion Criteria:

* A. Emergency Surgery for non-metastatic colorectal cancer B. Subjects who are being treated for recurrent colorectal cancer C. Subjects who will require extensive dissection to release adhesions or with advanced cancer which may result in anastomotic leak and/or bleeding unrelated to the stapler D. Subjects who have perforated, obstructing or locally invasive neoplasm (T4b) E. Subjects who have major concomitant abdominal or pelvic procedures (e.g. hepatectomies, incisional ventral hernia repair, nephrectomies, hysterectomy) planned along with surgery for colorectal cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rates | 24 MONTHS
  • Technological performance of stapler- Angle of stapler fire, Percent of cases with firing rate >45 degrees, Utility of AI Enabled (Smartfire) decision making- Clamp rates, fire rates

SECONDARY OUTCOMES:
Operative time | 24 MONTHS
  Operative time is defined as the total duration of the surgical procedure, measured in minutes, from skin incision to completion of skin closure.

CONTACTS AND LOCATIONS:
Overall Officials: DR G V RAO, MBBS,MAMS,FRCS, Principal Investigator — Asian Institute Of Gastroenterology Private Limited

IPD SHARING:
Plan to Share IPD: No